CLINICAL TRIAL: NCT06502418
Title: Impact of Acupuncture on Pain Management During Induced Labor with Cook's Balloon At the Beaumont Maternity in Roubaix
Brief Title: Acupuncture to Managed Pain During Induced Labor with Cook's Balloon
Acronym: COOKACUPAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Roubaix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-008
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Labor Induction
Keywords: Acupuncture therapy; Labor induction; Pain management
MeSH Terms: conditions — Agnosia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture arm (Experimental): Acupuncture therapy
  Interventions: Other: Acupuncture therapy
- Control arm (No Intervention): usual care

INTERVENTIONS:
Other: Acupuncture therapy — 7 acupuncture points will be used to managed pain and improved patient's experience
  Arms: Acupuncture arm

SUMMARY:
In France, labor induction rate is above 25.8%. Labor induction with Cook's balloon is a non-hormonal mechanical method but this technique can provide pain.

At Roubaix's maternity, midewifes can adminitred acupuncture therapy to help to manage this pain.

No studies where found about an effect of acupuncture therapy on pain provoked by labor induction with Cook's balloon.

DETAILED DESCRIPTION:
Investigators aim to demonstate that acupuncture therapy during labor induction with Cook's balloon can reduced pain and improved patient's experience. Investigators will use 7 acupuncture points (YIN TANG/ 4 GI bilateral/ 36 E bilateral and 5TR bilateral) before the application of the balloon. A visual analog scale will be used before and after balloon insertion to collect pain level.

a questionnary will be filled by patient to collect their experiences. Investigators will collect data about analgesia, failed of induction and cesarean section to see effect of acupuncture on them.

Patients will be randomised.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman with a gestational age of 37 weeks and above
* age>=18 years old
* having medical indication to be labor induced by Cook's Balloon
* speaking French
* agreeing to participate by signing informed consent form

Exclusion Criteria:

* patient having contraindication for the use of Cook's balloon
* patients under curatorship and/or guardianship

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Impact of 7 acupuncture points on pain | Day 1
  Assessment of pain with Visual Analogic Scale before and after the use of Cook's balloon

SECONDARY OUTCOMES:
Evaluate the consumption of analgesics between the 2 groups | Day 1
  datas of analgesics consumption will be collected in patient record
Evaluate experiences of the patient during labor induction between the 2 groups | Day 1
  Use of questionnary
Comparison of cesarean section rate, balloon failure rate and induction duration between the two groups | Day 2
  datas will be collected in patient record

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Roubaix, Roubaix, France